CLINICAL TRIAL: NCT02796742
Title: Prevalence of S. Aureus Among Patients Presenting With Skin and Soft Tissue Infections: a Multi-centre Pilot Study in Europe
Brief Title: S. Aureus, Skin and Soft Tissue Infections
Acronym: SSTIs
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0338
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Skin and Soft Tissue Infections (SSTIs)
Keywords: SSTIs; Methicillin-resistant Staphylococcus aureus (MRSA); Methicillin susceptible Staphylococcus aureus (MSSA); the toxin Panton-Valentine Leukocidin (PVL); Emergency Departments
MeSH Terms: conditions — Soft Tissue Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group MSSA
  Interventions: Other: Collecting samples from all patients presenting with SSTIs requiring drainage
- Group MRSA
  Interventions: Other: Collecting samples from all patients presenting with SSTIs requiring drainage
- Group PVL-negative strains
  Interventions: Other: Collecting samples from all patients presenting with SSTIs requiring drainage
- Group PVL-positive strains
  Interventions: Other: Collecting samples from all patients presenting with SSTIs requiring drainage

INTERVENTIONS:
Other: Collecting samples from all patients presenting with SSTIs requiring drainage — The study will be conducted by microbiology laboratories. Before the start of the study, each participating laboratory will send an information letter to its corresponding emergency departments to increase vigilance of clinicians in collecting samples from all patients presenting with SSTIs; this will improve the level of inclusion. Each participating lab will also insure connection to local representation of the project for ethical clearance, collection of clinical data and SSTI specimen.

SUMMARY:
Methicillin-resistant Staphylococcus aureus (MRSA) is reported as one of the main causative pathogen of community acquired SSTIs. In the USA, high prevalence of MRSA among Skin and soft tissue infections (SSTIs) is known to be due to the spread of the USA300 clone [Moran et al. 2006]. Among S. aureus SSTIs infections in Europe, data regarding the prevalence of MRSA in SSTIs and the causative genotypes remain scarce. The paucity of literature on the prevalence of MSSA, MRSA and PVL-producing S. aureus strains in SSTI in Europe is probably due to the fact that culture and antimicrobial susceptibility testing is not a routine component of SSTI management.

Setting-up a prospective multi-centre study involving patients presenting to emergency departments with SSTIs in several European countries would allow drawing a picture on the role and the respective contribution of MSSA, MRSA and PVL-producing S. aureus strains as a cause of SSTIs. However, the roles of emergency rooms and local policies with regard to performing microbiological analysis after surgical drainage of SSTIs vary between countries.

In order to evaluate the feasibility of such multicenter European study, we aim at performing a pilot study based on few European clinical laboratories (five to seven) which will: i) evaluate the prevalence of MSSA, MRSA and S. aureus PVL-positive strains in community-acquired SSTIs; and ii) determine molecular characteristics of the isolated strains. The main objectives of this pilot study are to collect some preliminary information on the role of S. aureus in SSTIs and to determine factors that need to be harmonized or taken into consideration for the set-up a larger prospective cross-sectional study involving more European countries with several centers per country to cover different geographical areas per country.

ELIGIBILITY:
Inclusion Criteria:

- All patients (adults and children) presenting to emergency department with purulent skin and soft tissue infections (SSTIs) of less than one week duration are eligible

Exclusion Criteria:

- Patients (adults and children) presenting to emergency department with OTHERS type of infections than SSTIs

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (adults and children) presenting to emergency department with purulent skin and soft tissue infections (SSTIs) of less than one week duration are eligible
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of staphylococcus aureus strains among all clinical SSTIs collected during the study. | after a 3 month period

SECONDARY OUTCOMES:
Percentage of MSSA, MRSA strains among all clinical SSTIs collected during the study | after a 3 month period
Percentage of PVL-positive strains among all clinical SSTIs collected during the study | after a 3 month period

CONTACTS AND LOCATIONS:
Overall Officials: François Vandenesch, Pr, Principal Investigator — National Reference Center for Staphylococci
Locations (1):
- National Reference Center for Staphylococci, 59 boulevard Pinel, Bron, France

REFERENCES:
- [Background] Moran GJ, Krishnadasan A, Gorwitz RJ, Fosheim GE, McDougal LK, Carey RB, Talan DA; EMERGEncy ID Net Study Group. Methicillin-resistant S. aureus infections among patients in the emergency department. N Engl J Med. 2006 Aug 17;355(7):666-74. doi: 10.1056/NEJMoa055356. PMID 16914702